CLINICAL TRIAL: NCT03331302
Title: Hyper Polarized Xenon-129 MRI vs Xenon-133 Scintigraphy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Associate Professor, University of Virginia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 20053
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pilot Projects

STUDY DESIGN:
Intervention Model Description: COPD patients with standard vs study diagnostic methods (imaging procedures)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COPD patients - Xe-133 (Active Comparator): COPD patients who will be assessed with Xenon-133 scintigraphy (Standard diagnostic study)
  Interventions: Drug: Radioactive Xenon-133 scintigraphy (Active Comparator)
- COPD patients - Hyperpolarized Xe-129 (Experimental): COPD patients crossed over from the Active Comparator Arm who will be assessed with hyper polarized Xenon-129 MRI (Experimental diagnostic study)
  Interventions: Drug: Hyperpolarized Xenon-129 MRI (Experimental)

INTERVENTIONS:
Drug: Hyperpolarized Xenon-129 MRI (Experimental) — MRI ventilation scan of the lung with inhaled contrast agent (hyperpolarized Xenon-129)
  Other Names: Polarean Pilot study
  Arms: COPD patients - Hyperpolarized Xe-129
Drug: Radioactive Xenon-133 scintigraphy (Active Comparator) — Radioactive ventilation scintigraphy of the lung with inhaled radioactive contrast agent (Xenon-133)
  Other Names: Pilot study
  Arms: COPD patients - Xe-133

SUMMARY:
Hyper polarized Xenon-129 MRI will be directly compared to a radioactive Xe-133 scintigraphy to detect defects in lung ventilation from airflow limitation. This study is conducted as a pilot study with intention to conduct a larger clinical trial.

DETAILED DESCRIPTION:
Hyperpolarized Xenon-129 MRI has been developed by a number of techniques for imaging the lung that provide information about various aspects of lung function and structure. The main objective of this pilot study is to test and optimize the imaging parameters for a future industry sponsored clinical trial. The goal of the future trial is to determine the concordance between hyperpolarized xenon-129 ventilation MR imaging and nuclear medicine ventilation imaging (Gold Standard). In this study we will test the imaging parameters and techniques. We will directly compare human ventilation lung images in subjects with COPD, using nuclear medicine ventilation imaging with Xenon-133 gas scintigraphy versus hyperpolarized xenon-129 gas MRI. Our hypothesis is that current Xe-133 scintigraphy, which uses a radioactive gas (Xe-133) and produces a projection image of the lungs with relatively poor resolution, will not be able to detect small lung ventilation obstructions, which can be detected using hyperpolarized Xe-129 gas MRI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of COPD
* at their clinical baseline on the day of imaging
* must be clinically stable in order to participate in the study.
* COPD subjects will be categorized according to the GOLD
* Current/Former SmokerSubjects
* must have a smoking history ≥ 10 pack years

Exclusion Criteria:

* Dx of asthma
* Continuous oxygen use at home
* Blood oxygen saturation of 92% less than as measured by pulse oximetry on the day of imaging
* FEV1 percent predicted less than 25%
* Pregnancy or lactation
* Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in eye, pacemaker or other contraindication to MR scanning
* Subjects with any implanted device that cannot be verified as MRI compliant will be excluded
* Chest circumference greater than that of the xenon MR and/or helium coil. The circumference of the coil is approximately 42 inches
* History of congenital cardiac disease, chronic renal failure, or cirrhosis
* Inability to understand simple instructions or to hold still for approximately 10 seconds
* History of respiratory infection within 2 weeks prior to the MR scan
* History of MI, stroke and/or poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventilation imaging resolution comparison between MRI and scintigraphy | 12 months
  Compare the quality of the imaging between hyper polarized xenon-129 and radioactive xenon-133

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided for now.